CLINICAL TRIAL: NCT06581666
Title: Current Awareness, Perspective and Knowledge on Social Egg Freezing
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2024.346
Record Dates: First submitted 2024-08-22; First posted 2024-09-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All patients who have undergone or will seek fertility preservation services: All patients who have undergone or will seek fertility preservation services, but they will be asked to complete the same set of questionnaires.
  Interventions: Other: No special intervention, all participants will be asked to complete same set of questionnaire.
- General public: The general public will also be asked to complete the sane set of questionnaires.
  Interventions: Other: No special intervention, all participants will be asked to complete same set of questionnaire.

INTERVENTIONS:
Other: No special intervention, all participants will be asked to complete same set of questionnaire. — No special intervention, all participants will be asked to complete same set of questionnaire.

SUMMARY:
Hong Kong's fertility preservation service is underutilized and limited, with low awareness among clinicians and young adults. Traditional Chinese culture may lead to social stigma, preventing discussion of fertility issues. A survey aims to explore awareness, knowledge, and acceptance of oocyte cryopreservation, enabling resource allocation for a culturally acceptable public education program and a dedicated referral system to improve oocyte cryopreservation services.

DETAILED DESCRIPTION:
Hong Kong's fertility preservation service is underutilized and limited, with low awareness among clinicians and young adults. Traditional Chinese culture may lead to social stigma, preventing discussion of fertility issues. A survey aims to explore awareness, knowledge, and acceptance of oocyte cryopreservation, enabling resource allocation for a culturally acceptable public education program and a dedicated referral system to improve oocyte cryopreservation services.

The questionnaire will be in paper form and as an online survey. Potential participants will be provided with the study aim and respondent rights. Once verbal informed consent is obtained, participants will be asked to fill in the self-administered questionnaire. For the online survey, implied consent from the participants will be adopted when they complete the questionnaire on the webpage and return it to us.

In order to reach the 2 target groups, convenient sampling will be used. Questionnaires will be distributed to the patients who have undergone or will seek fertility preservation services in PWH. For the general public, they will be recruited online via an invitation link.

ELIGIBILITY:
Inclusion Criteria:

* People with aged from 18-60 years old

Exclusion Criteria:

* Patients unable to provide consent/assent (i.e. significant psychiatric problems/cognitive delay)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients aged from 18-60 years old, who have undergone or will seek fertility preservation services in PWH and the general public will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Awareness, perspective and knowledge | through study completion, an average of 1 year
  To evaluate the difference in the level of awareness, perspective and knowledge towards social egg freezing between patients who have undergone or will seek fertility preservation services and the general public.

SECONDARY OUTCOMES:
Awareness | through study completion, an average of 1 year
  To evaluate the awareness of oocyte cryopreservation among the general public and patients
Factors that may affect the uptake rate | through study completion, an average of 1 year
  To determine any factors that may affect the uptake rate of oocyte cryopreservation
Utilization rate | through study completion, an average of 1 year
  To assess the utilization rate of social egg freezing

CONTACTS AND LOCATIONS:
Overall Officials: PUI WAH JACQUELINE CHUNG, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Pui Wah Jacqueline Chung, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No